CLINICAL TRIAL: NCT00819650
Title: Eastern Hepatobiliary Surgical Hospital
Brief Title: A Trial of Licartin for Preventing Tumor Recurrence After Liver Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-014-1
Record Dates: First submitted 2009-01-01; First posted 2009-01-09 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; adjuvant therapy; Licartin; time to recurrence; overall survival
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — metuximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Licartin (Experimental): patients who receive Licartin therapy after liver resection
  Interventions: Drug: Licartin (generic name,[131I]metuximab injection)
- placebo (No Intervention): control group with patients who don't receive any adjuvant therapy after liver resection, to compare with the treatment group with patients who receive Licartin therapy after liver resection

INTERVENTIONS:
Drug: Licartin (generic name,[131I]metuximab injection) — Licartin, radioiodination of Metuximab with Na[131I],with radiochemical purity above 95% and specific activity between 173.25-288.75 MBq/ml.All patients in the treatment group received Licartin 3 times at an interval of 28 days beginning from the 4th week after liver resection
  Other Names: no adjuvant therapy after liver resection
  Arms: Licartin

SUMMARY:
The aim of this study is to analyze the therapeutic effect of adjuvant Licartin therapy after resection.Patients receiving curative resection (R0) were randomized to postoperative Licartin group and no Licartin group. The time to recurrence ,the overall survival as well as the incidence of complications after therapy was observed to confirm the role of adjuvant therapy of Licartin.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) represents a major health care challenge in the present era, with its incidence rate of 71128 cases and the mortality rate of 679871 cases during 2007 in the world. Although liver transplantation, resection and locally ablative therapies remain useful treatment preference in patients with early HCC, but they often cannot be availed because of either disease progression or outgrowth of treatment criteria, especially for liver resection. Moreover, after resection, recurrence of liver tumor can be expected in as many as 70% of patients within 5 years which leading to the unsatisfactory long term survival of patients with HCC, hence prevention and effective management of recurrence are undoubtedly the major strategies to prolong the survival. And until now although a lot of different adjuvant therapies had been tried in the clinic, including TACE, immunotherapy and antivirus therapy etc. their role in preventing recurrence remain controversial.

Licartin (generic name, [131I]metuximab injection), a member of CD147 family and a therapeutical anti-HCC radioimmunologic agent, generated by labeling of 131I with murine monoclonal antibody (mAb) target fragment HAb18 F(ab_)2, was approved as a new drug for clinical therapy of primary HCC by China State Food and Drug Administration for its good concentrate in the tumor region and safe and effective treatment of HCC. Previous RCT study indicated that Licartin prevented post-Orthotopic liver transplantation(OLT) tumor recurrence in advanced HCC patients exceed Milan criteria. The recurrence rate significantly decreasing by 30.4% at 1-year follow up in the OLT group compared with those in the control group showed that Licartin may be a promising drug for preventing tumor recurrence after liver transplantation. But less information is known about its role as an adjuvant therapeutic drug after liver resection. To determine the clinical efficacy of Licartin for preventing tumor recurrence after liver resection, we set up a randomized, controlled trial in patients who were definitely diagnosed with HCC and who were successfully treated with liver resection.

Patients with HCC who received curative liver resection (R0)and with positive expression of HAb18G/CD147 in the HCC tissues were randomly assigned 1:1 by the doctors to receive placebo(control group) or Licartin (treatment group). All patients in the treatment group received Licartin 3 times at an interval of 28 days beginning from the 4th week after liver resection. The outcomes of patients were evaluated during the 3-years follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with HCC who received curative liver resection (R0)and with positive expression of HAb18G/CD147 in the HCC tissues
2. Karnofsky Performance Score performance over 60
3. The functions of the kidney, heart and lung and the blood system are normal and fittable for Licardin therapy.
4. The liver function is of grade A or B in Child-Pugh classification.
5. Patients give consent to the test.

Exclusion Criteria:

1. Negative expression of HAb18G/CD147 in the HCC tissues
2. Allergic history to biologic products(Licartin)
3. Any of the situation list below: WBC less than 2000/ml, Hb less than 90g/L or PLT less than 50000/ml, bilirubin level more than 2.5 times the upper limit of normal value, serum albumin less than 32 g/l.
4. Severed disease of the heart, lung, kidney, brain and blood system.
5. Other severed disease might affect the trial .
6. Patients would not sign the consent to the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2010

SECONDARY OUTCOMES:
Time to recurrence | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, MD, Study Chair — Eastern hepatobilliary surgery hospital
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li J, Xing J, Yang Y, Liu J, Wang W, Xia Y, Yan Z, Wang K, Wu D, Wu L, Wan X, Yang T, Gao C, Si A, Wang H, Wu M, Lau WY, Chen Z, Shen F. Adjuvant 131I-metuximab for hepatocellular carcinoma after liver resection: a randomised, controlled, multicentre, open-label, phase 2 trial. Lancet Gastroenterol Hepatol. 2020 Jun;5(6):548-560. doi: 10.1016/S2468-1253(19)30422-4. Epub 2020 Mar 9. PMID 32164877